CLINICAL TRIAL: NCT00017134
Title: An Exploratory Evaluation of Fenretinide (4-HPR) as a Chemopreventive Agent for Ovarian Carcinoma
Brief Title: Fenretinide Followed by Surgery Compared With Surgery Alone in Preventing Ovarian Cancer in Patients at Increased Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to poor accrual
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000068655; GOG-0190
Record Dates: First submitted 2001-06-06; First posted 2003-05-07 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2006-11

CONDITIONS: Ovarian Cancer
Keywords: ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Fenretinide

INTERVENTIONS:
Drug: fenretinide
Procedure: conventional surgery

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer. It is not yet known whether fenretinide given before surgery is more effective in preventing ovarian cancer than surgery alone.

PURPOSE: Randomized clinical trial to compare the effectiveness of fenretinide followed by surgery with that of surgery alone in preventing ovarian cancer in patients who are at increased risk.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the frequency of histopathology markers or precursor lesions of the ovaries, including surface papillomatosis, invaginations, pseudostratification, and inclusion cysts, removed from patients at increased risk for ovarian cancer between those receiving fenretinide vs those undergoing immediate oophorectomy.
* Determine the relative abundance of markers of cell proliferation and apoptosis in cancer-prone ovaries of patients treated with fenretinide.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 arms.

* Arm I: Patients undergo prophylactic oophorectomy.
* Arm II: Patients receive oral fenretinide once daily for 27 days every 30 days for 6-8 weeks. Treatment continues in the absence of unacceptable toxicity or diagnosis of malignancy. After completion of fenretinide, patients undergo prophylactic oophorectomy.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 71 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Increased risk for ovarian cancer secondary to 1 of the following:

  * Evidence of a BRCA1 or BRCA2 genetic mutation
  * Family history of 1 or more first-degree relatives diagnosed with ovarian cancer prior to 50 years of age
  * Family history of 1 first-degree relative with ovarian cancer (any age) AND 1 or more first- or second-degree relatives diagnosed with breast or ovarian cancer
  * Personal history of breast cancer (at any age) AND 1 or more first- or second-degree relative diagnosed with breast or ovarian cancer at any age
* Meets any 1 of the following criteria:

  * Ashkenazi Jewish ethnicity with 1 first-degree or 2 second-degree relatives with breast* and/or ovarian cancer
  * Ashkenazi Jewish ethnicity with diagnosed breast* cancer in patient
  * Greater than 20% probability of carrying BRCA1/2 mutation with a family history of breast and ovarian cancer NOTE: * Where breast cancer is required to meet this criteria, diagnosis must occur prior to menopause or at ≤ 50 years old if age at menopause is unknown
* Planned prophylactic oophorectomy
* Normal pelvic exam within the past 6 weeks

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* GOG 0-1

Life expectancy:

* At least 12 months

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* Triglyceride less than 2 times ULN (fasting)

Cardiovascular:

* No myocardial infarction within the past 3 months
* No active angina
* No unstable heart rhythms
* No clinically evident congestive heart failure

Other:

* No uncontrolled medical illness that would preclude study participation
* No uncontrolled diabetes
* No uncontrolled psychiatric illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 months since prior chemotherapy

Endocrine therapy:

* At least 3 months since prior hormonal therapy
* At least 8 weeks since prior hormone replacement therapy
* At least 8 weeks since prior oral, injectable, or implantable contraceptives
* No concurrent hormonal therapy, including hormone replacement therapy

Radiotherapy:

* At least 3 months since prior radiotherapy
* No prior radiotherapy to pelvis for malignancy

Surgery:

* See Disease Characteristics

Other:

* At least 3 months since prior investigational treatment
* No concurrent nutritional supplements except a daily multivitamin with less than 25,000 IU of vitamin A
* No prior non-steroidal anti-inflammatory drugs (NSAIDs) on a regular (chronic or daily) basis within the past 6 months
* No concurrent NSAIDs on a regular (chronic or daily) basis
* Concurrent aspirin at a dose of 81 mg/day allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2002-09; Primary Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary B. Daly, MD, PhD, Study Chair — Fox Chase Cancer Center
Locations (35):
- United States (35):
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Colorado Gynecologic Oncology Group P.C., Aurora, Colorado
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - George Bray Cancer Center at New Britain General Hospital, New Britain, Connecticut
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - University of Minnesota Medical Center & Children's Hospital - Fairview, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia